CLINICAL TRIAL: NCT01531335
Title: Effectiveness of Hypocaloric Nutrition Compared With Standard Care in Critically Ill Adults Patients, a Randomized Controlled Trial
Brief Title: Hypocaloric Nutrition in Critically Ill Patients
Acronym: RuRaL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lafrancol S.A. (Industry)
Collaborators: Hospital Universitario San Ignacio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SJ0079
Record Dates: First submitted 2012-02-07; First posted 2012-02-10 (Estimated); Results first posted 2015-12-11 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-11

CONDITIONS: Critically Ill
Keywords: adults
MeSH Terms: conditions — Critical Illness | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard care (Active Comparator): Patients will receive normal nutritional regime of around 25 kcal per kg.
  Interventions: Dietary Supplement: Standard care
- Hypocaloric hyperproteic nutrition (Experimental): 15 kcal per kg of body weight and 1.7 grams of protein per kg
  Interventions: Dietary Supplement: Hypocaloric hyperproteic nutrition

INTERVENTIONS:
Dietary Supplement: Hypocaloric hyperproteic nutrition — 15 kcal per kg of body weight and 1.7 grams of protein per kg.
  Other Names: Hypocaloric hyperproteic
  Arms: Hypocaloric hyperproteic nutrition
Dietary Supplement: Standard care — 25 kcal per kg of body weight
  Other Names: Isocaloric
  Arms: Standard care

SUMMARY:
The aim of this study is to compare two nutritional regimes in critically ill patients. Patients will be randomized to standard care (25 kcal per kg) or to hypocaloric nutrition (15 kcal per kg). The main outcome will be the SOFA (sequential organ failure assessment) score. The hypothesis is that hypocaloric hyperproteic diet decreases the incidence of organic failure in these patients.

DETAILED DESCRIPTION:
The research site will be the intensive care unit (ICU) of Hospital Universitario San Ignacio; eligible patients will >18 years of age with a presumed fasting period of at least 96 hours, with no contraindications for enteral nutrition. Patients with parenteral nutrition, pregnancy, diabetes, liver failure, renal failure, transplant protocol, or admitted from another hospital will be excluded. In all patients, the following information will be collected daily: enteral formula in ml, carbohydrate intake, insulin required (in IU), presence of hyper or hypoglicemia, presence of infections, among others.

The SOFA score will be assessed every two days until discharge from ICU.

ELIGIBILITY:
Inclusion Criteria:

* >18 years
* estimated fasting period of at least 96 hours

Exclusion Criteria:

* parenteral nutrition
* pregnancy
* diabetes
* liver or renal failure
* transplantation
* admitted from another hospital

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2011-08; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saul Rugeles, MD, Principal Investigator — Pontificia Universidad Javeriana
Locations (1):
- Hospital Universitario San Ignacio, Bogotá, DC, Colombia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Care | Hypocaloric Hyperproteic Nutrition
Started | 40 | 40
Completed | 40 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Care | Hypocaloric Hyperproteic Nutrition | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.7 (19.5) | 53.3 (19.5) | 54.5 (19.5)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 40 | 40 | 80
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 18 | 34
  Male | 24 | 22 | 46
Region of Enrollment [Number; unit: participants]
  Colombia | 40 | 40 | 80

OUTCOME MEASURES:

1. Primary Outcome: SOFA (Sequential Organ Failure Assessment) Score
Description: SOFA score evaluates six systems: respiratory, cardiovascular, coagulation, Central Nervous System, liver and renal. Each system gets a score from 0 (normal) to 4 (abnormal) and the sum of each score defines the final SOFA score, which 24 is the maximum score (high risk of morality) and 0 is the minimum score (low risk of mortality).
Time Frame: 48 hours since nutritional regime starts
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Care | Hypocaloric Hyperproteic Nutrition
Number analyzed (Participants) | 40 | 40
units on a scale | 0.7 (2.8) | 1.7 (1.9)

2. Secondary Outcome: Insulin Requirements
Description: This is an indirect measure of glycemic control, and is reported as a daily average.
Time Frame: Daily until day 21 or discharge from ICU
Measure: Mean (Standard Deviation); unit: International Unit of insulin
Arm/Group | Standard Care | Hypocaloric Hyperproteic Nutrition
Number analyzed (Participants) | 40 | 40
International Unit of insulin | 14 (22.1) | 10.4 (17.8)

ADVERSE EVENTS:
Arm/Group | Standard Care | Hypocaloric Hyperproteic Nutrition
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

LIMITATIONS AND CAVEATS:
No surgical patients included Wide variety of patients Caloric needs were not estimated with a gold standard

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No